CLINICAL TRIAL: NCT06091163
Title: A Randomised Controlled Trial Evaluating the Efficacy and Mechanisms of a Ketogenic Diet as an Adjunctive Treatment for People With Treatment-resistant Depression
Brief Title: Ketogenic Diet for Treatment-Resistant Depression: Dietary Interventions for MEntal Health Study (DIME)
Acronym: DIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Sheffield (Other); McPin Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R87397
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Treatment Resistant Depression; Depression; Mental Illness; Mental Disorder; Depressive Disorder
Keywords: Ketogenic Diet; Keto Diet; Keto; Metabolic Ketosis; Randomised Controlled Trial
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Mental Disorders; Depressive Disorder; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (KD) (Experimental): Participants allocated to this condition will receive 6-weeks of home-delivered pre-prepared ketogenic diet (KD) meals (3 meals/day, snacks) from a vetted ketogenic diet food supplier. The 6-week intervention includes a weekly 30-minute dietary counselling call with a registered dietitian to support following a ketogenic diet. Participants receive educational materials with information about foods that are compatible with the diet, common symptoms and how to manage them, and strategies to help maintain the diet during and after the 6-week intervention period.
  Interventions: Behavioral: Ketogenic Diet
- Phytonutrient Diet (PD) (Placebo Comparator): Participants in the control group will receive weekly 30-minute dietary counselling with a registered dietitian and be asked to increase vegetable consumption and reduce saturated fat intake as part of a phytonutrient diet (PD). Participants will receive food vouchers every 2-weeks to help purchase food items or replacements that support high vegetable, low saturated fat intake. This aims to be a plausible placebo dietary treatment for depression. There is no clear evidence that these manipulations will change depression severity. The dietitian will provide materials to explain the diet and suggest foods by colour with supporting recipe suggestions.
  Interventions: Behavioral: Phytonutrient Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — A Ketogenic Diet (KD) is a high-fat and very low-carbohydrate intake. Participants will follow a modified KD (estimated 20-50g carbohydrates/day based on a 2000 kcal diet) without energy restriction. Participants will test for ketosis in their morning urine at least twice a week to monitor adherence.
  To support adherence in people with depression, delivered pre-prepared KD meals (3 meals per day) and additional ketogenic snacks will be sent to participants. A registered dietitian will provide weekly 30-minute nutritional counselling sessions. The dietitian will schedule appointments and assess the participants' experience with adhering to the KD diet, troubleshoot as required, give guidance on how to prevent or overcome side effects of KD diets, and keep record of participants' ketosis level and suicide risk.
  Other Names: Keto Diet
  Arms: Ketogenic Diet (KD)
Behavioral: Phytonutrient Diet — Participants in the control group will receive the same degree of dietetic input and be told that their diet is a modified fat and phytonutrient diet. The photo diet aims to increase vegetable consumption, reduce saturated fat intake and increase poly- and mono-unsaturated fat intake. Participants in the control group will receive food vouchers (£20 every two weeks) to help purchase these items. This aims to be a plausible placebo dietary treatment for depression. There is no clear evidence that these manipulations will change depression severity. The dietitian will create written materials to explain the diet and suggest foods by colour with supporting recipe suggestions.
  Other Names: Phyto Diet
  Arms: Phytonutrient Diet (PD)

SUMMARY:
Depression is a debilitating chronic illness affecting 1 in 6 adults in the United Kingdom (UK) at any one time. Antidepressants and psychological therapy are the main treatments, but some people do not respond to these. Neurons and signals in the brain are greatly disrupted in people with severe depression. A ketogenic diet, a high-fat and very low-carbohydrate diet, supplies a form of energy that appears to help brain cells communicate and may improve the treatment of depression. Our goal is to find out whether a ketogenic diet could be an additional effective treatment for patients with depression for which antidepressants do not work.

Using social media advertising, 100 patients, ages 18-65, who have previously tried at least two different antidepressant medications within the current depressive episode will be recruited. Enrolment, consent, and data collection will be collected online using self-report questionnaires. Participants will be allocated by minimisation 1:1 to the KD group or control group based on depressive severity (moderately severe vs. severe) and body mass index (<30kg/m2 vs. 30+ kg/m2). The intervention group will receive 6-weeks of prepared ketogenic diet meals (3 meals with snacks per day) and weekly ketogenic diet-focused nutrition counselling. The control group will be asked to follow a diet to reduce their saturated fat intake and increase vegetable consumption by one portion a day. The control group will receive vouchers to assist with purchases and will be provided with weekly nutritional counselling. Existing treatment for depression will remain in both groups.

The primary outcome is the change in depression symptoms at six weeks. All participants will complete assessments of depression and anxiety every two weeks, starting before treatment to post-intervention (week 6), and again at week 12. Additional outcomes include participants' ability to experience pleasure, quality of life, ability to socialise and work, cognitive processing, morning cortisol, and gut microbiome.

At all stages of the study, adults with lived experience of depression will advise the research team to take into account the needs and views of patients.

This study will provide evidence of whether following a ketogenic diet leads to a short-term improvement in depression in people whose depression cannot be relieved by antidepressants.

DETAILED DESCRIPTION:
One in 6 people suffer from clinical depression. Antidepressants are a first-line treatment for depression, but at least 1 in 3 patients with depression do not respond to antidepressants and not everyone responds to, or wants psychological therapy. Furthermore, there is still a high relapse rate after psychological treatment. Longer depressive episodes, a higher number of hospitalisations, moderate to high suicide risk, physical and psychiatric comorbidities, and higher dosage of medication, were partly explained by the low response (16-17%) and remission rates (13%). Hence, new treatment options for treatment resistant depression (TRD) are needed.

Recent research in depression indicates that the imbalance between excitatory (e.g. glutamatergic system) and inhibitory (e.g. GABA system) systems may be a better way of understanding depression. There is strong evidence that GABAergic neurotransmission is disrupted in depression and concentrations of GABA are significantly reduced, especially in treatment-resistant depression. This suggests increasing inhibitory neurotransmitters (e.g. GABA) could be an alternative way to treat depression.

KDs (ketogenic diets), characterised by high-fat and very low-carbohydrate intake, have been recently suggested as a possible intervention for depression due to the influence on neurotransmitters. KDs increase production of the inhibitory neurotransmitter GABA, and restore microglial activation and neuronal excitability in the lateral habenula, a region involved in negative reward processing. Furthermore, the mechanisms of action of KD appear to include several additional potential mechanisms of action in depression including cellular bioenergetics, reduced oxidative stress, improved brain vascularity, and influence on the HPA axis (via lowered cortisol), and changes in gut microbiome.

Despite several plausible beneficial effects and increased public interest and rapid market growth of KD food products (estimated $12.4 billion by 2024), and evidence of biological plausibility demonstrated in epilepsy and animal models, the efficacy of KDs for treatment-resistant depression has not yet been established. To our knowledge, there are only three registered clinical trials underway testing KD for mental disorders, however, none examine efficacy of KD for treatment-resistant depression and there are no currently published results. A recent systematic review is the first to appraise the literature on KD for mental disorders in human samples and highlights the paucity of robust research. Twelve studies examining 388 participants (9 case reports, 2 cohort studies, and one observational study) met inclusion criteria and found no high-quality evidence of KD efficacy for mental disorders. The absence of controlled trials, heavy reliance on individual case studies, grouping of various clinical disorders together, lack of uniform definition of KD across studies, including five studies not reporting KD nutritional intake, and no measurement of ketosis in half the studies make interpretation of the literature difficult. However, the review data suggest that people with various mental illnesses who follow a KD can have marked improvements in mental health. Moreover, a recent review suggests that symptom scales such as the PHQ-9 may be useful but should be better combined with measures of functioning and quality of life to fulfil patients' perspectives.

The current study proposes to test whether a 6-week ketogenic diet is an effective treatment for treatment-resistant depression. Recruitment of 100 participants with treatment-resistant depression based on a sample size calculation will be conducted. A 5-point difference in PHQ-9 will be considered to represent a clinically important difference based on prior research. This study reported that the Standard Deviation (SD) of the change in PHQ-9 over 3 months as 5.8 and as 6.1 over 6 months. Assuming an SD of 6 over 6 weeks would suggest a standardised effect size of 0.83 in PHQ-9 to be clinically relevant. The sample size to test differences between groups at 90% power and at a type one error rate of 5% would be 64 (32 per group). A sample size of 100 participants will be recruited to make the study robust against up to 35% attrition/missing data. In simulations, it has been confirmed that this sample size remains robust under scenarios such as unequal sizes of the strata used in minimisation.

After all baseline assessments are complete, participants will be allocated by minimisation 1:1 to the KD group or control group. A researcher will embed a non-deterministic algorithm in the Redcap database. This algorithm aims to produce treatment groups balanced for important prognostic factors by minimising on the following variables (as below). Only after eligibility and consent is confirmed will the database reveal the allocation. Investigators delivering the intervention will not be blinded, but the outcome is collected blind (by self-report), and those involved in analysing the outcome data will be blinded to allocation.

* BMI (less than 30 kg/m2 vs. 30+ kg/m2)
* Depression severity (PHQ-9 score: 15-19 [moderately severe] vs. 20-27 [severe])

All follow-up is done online and without trial staff and will therefore not be subject to observation bias.

Following randomisation, participants will be given information and advice for their respective group. The KD group involves 6-week pre-prepared ketogenic diet with weekly KD-focused behavioural and nutritional counselling. The control group will receive weekly nutritional counselling to increase vegetable consumption and reduce saturated fat intake. Participants in the control group will receive food vouchers to help purchase these items. This aims to be a plausible placebo dietary treatment for depression. Usual treatment for depression will continue, and leaflet material is provided in both groups.

Psychometric questionnaires and biological outcomes will be assessed pre-post intervention, and at 12-week follow-up, to investigate changes in depression symptom severity and potential mechanistic pathways.

Initial descriptive statistics will present the profile of the subjects by study arm without using statistical comparisons. For the primary hypothesis, the change in PHQ-9 scores from baseline to week 6 will be compared between groups. A mixed effect model that includes treatment group, time and their interaction as fixed effects, and individual subjects as random effects will be fit using PHQ-9 at all available assessments. A linear contrast will be used to test the difference between groups in changes from baseline to week 6 in PHQ-9 scores. Two tailed tests and significance level of 0.05 will be used. Secondary outcomes will be analysed using analogous mixed effects generalised linear models. Pre-specified subgroup analyses of the primary outcome will be explored by baseline depression severity (severe versus moderate) and duration of depression at baseline split at the median. An exploratory mediation analysis using previously validated methods to examine whether adherence to the diet, changes in microbiome, and cortisol awakening response appear to mediate changes in depression. Spearman correlations will determine associations between alpha diversity metrics, individual microbes, and PHQ-9 scores. Kruskal-Wallis one-way analysis of variance tests will be performed to compare relative abundance of the top ten genera, with false discovery rate (FDR) corrections between dietary groups. Complete case analysis will be used as the primary analysis if the proportion of missing data is below 5%. A sensitivity analysis to explore reasons for missingness and determine appropriate handling of missing data will be conducted.

A 12-member advisory panel of adults with lived experience of mental and physical illness (50% from ethnic minority backgrounds) in collaboration with The McPin Foundation has been formed to inform all stages of this research trial. Members have expressed interest to know whether KDs can treat depression, and they welcome this kind of research. An additional 8 members of the public who have depression, of whom 3 had previously followed a KD diet were involved in the study design (e.g. social media and public advertising to engage participants, prepared meals preferred, motivational messages, strategies aimed at addressing relapsing and relapse following KD diets) before ethics submission. Participants in the trial will be offered the opportunity to hear the results of the study upon completion, and a lay summary and infographic will be provided.

A six-member trial steering committee (TSC) has been formed to provide independent oversight of the trial. Three independent members (50%) whose scientific, psychiatric, and statistical expertise is directly relevant to the trial, have verified they have no relationship to the investigators, the trial funders, nor employed by the same institution. The TSC will meet at least annually at appropriate time-points to ensure the trial is conducted in accordance with clinical trial standards.

There are few established and widely available treatments available for people with TRD. This is the first randomised, controlled trial assessing the effects of KDs on symptoms of depression in patients with TRD. Findings from this trial will provide evidence of efficacy of a new option for alleviating depressive symptoms in people who do not respond to antidepressants. If the treatment proves efficacious, it will create a potential new way to treat these patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Have been diagnosed with depression
* Currently on an antidepressant medication for a period of 4-weeks or longer
* Have tried 2 or more antidepressant treatment trials of adequate dose and duration within the current depressive episode to which they did not fully respond. An adequate treatment trial is defined as at least 4 weeks of a medication at a minimum National Institute for Health and Care Excellence (NICE) approved dose
* With a Patient Health Questionnaire-9 (PHQ-9) total score greater than or equal to 15 at baseline
* Able to understand and be willing to adhere to the demands of the study
* Provision of written informed consent
* Have access to a tablet/computer for online assessments, follow-ups with the registered dietitian, and able to attend appointments for assessments and treatment and adhere to study procedures
* Have both a fridge and a freezer at home
* Complete all baseline assessments

Exclusion Criteria:

* Currently following a low carbohydrate or ketogenic diet
* Currently following a vegan or vegetarian diet as these diets are more challenging to accommodate in a Ketogenic Diet and adding vegetables in the control group is unlikely to be seen as helpful.
* Currently receiving, or have received, in-patient psychiatric treatment or electroconvulsive therapy (electric shock to the brain under brief general anaesthetic) within the past year, or scheduled to receive such treatment during the study
* Currently using St John's wort or other remedies for depression that were bought without a doctor's prescription
* Currently have suicidal ideation with intent* or attempted suicide within the past two months
* Ever had an eating disorder, bipolar disorder, schizophrenia, or psychosis
* Have substance use or alcohol dependence
* Have epilepsy
* Have serious food allergies (experiencing food hypersensitivity that leads to anaphylaxis or other severe symptoms, which may require hospitalisation or are life-threatening) or otherwise require a special diet that cannot be accommodated within a KD such as phenylketonuria or lactose intolerance
* Treated with insulin, sulfonylureas, Glucagon-like peptide-1 (GLP-1) agonists, or Sodium-glucose co-transporter-2 (SGLT2) inhibitors
* Women who are pregnant, planning pregnancy in the next three months, or breastfeeding
* Have a body mass index (BMI) of <18.5 kg/m2
* Have unstable or severe medical conditions (e.g., cancer, cardiovascular, renal, lung, psychiatric, or bleeding disorders, diabetes, etc.), currently receiving cancer treatment except hormonal treatment for breast cancer or non-melanoma skin cancer treatment
* Have gallstones, renal tubular acidosis, kidney stones, small bowel malabsorption or a history of pancreatitis
* Have scheduled a major surgery in the next 3 months
* Taking part in other studies that may compromise this study or this study may compromise the other study/ies
* Have read the trial protocol or the clinical trial registration information and therefore are unblinded
* Live in the same household as another participant in the trial
* Not able to complete the online task with a tablet/computer
* Not willing to provide saliva, urine and stool samples

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline, 2 weeks, 4 weeks, 6 weeks (post-intervention), 12 weeks (follow-up)
  The PHQ-9 is a previously validated and reliably self-administered 9-item questionnaire of depression severity corresponding to Diagnostic Statistical Manual 5th Edition (DSM-V) criteria for major depressive disorder. Items are scored on a 4-point scale from "0" = not at all to "3" = nearly every day. Total scores range from 0 to 27 with higher scores reflecting increased depression severity. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
General Anxiety Disorder Scale (GAD-7) | Baseline, 2 weeks, 4 weeks, 6 weeks (post-intervention), 12 weeks (follow-up)
  The GAD-7 is a 7-item self-administered questionnaire measuring worry and anxiety symptoms. Items are scored on a 4-point Likert scale (0-3) with total scores ranging from 0 to 21. Higher scores indicate greater symptom severity of anxiety. Scores > 10 are indicative of clinical symptoms. The GAD-7 has shown previous reliability and construct validity.
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, 6 weeks (post-intervention), 12 weeks (follow-up)
  The SHAPS is a 14-item scale that measures the inability to experience pleasure (anhedonia). Items are rated on a 4-point Likert scale ranging from strongly disagree, disagree, agree, strongly agree. A score of 1 is given to either the disagree/strongly disagree responses, and a score of 0 is given to either the agree/strongly agree responses. Total scores range from 0 to 14 with higher scores reflecting greater anhedonia (inability to experience pleasure). The SHAPS has previously shown adequate validity and reliability, and high internal consistency.
Perceived deficits questionnaire-5-item (PDQ-5) | Baseline, 6 weeks (post-intervention), 12 weeks (follow-up)
  The PDQ-5 is a validated and reliable abbreviated, brief 5-item self-administered questionnaire to assess subjective cognitive dysfunction in people with depression. Items are rated on a 5-point scale of 0 = never to 4 (very often - more than once a day). Total scores for the PDQ-5 ranges from 0 to 20 with higher scores reflecting worse perceived cognitive deficits.
The Medical Outcomes Study (MOS) 12-item Short-Form Health Survey (SF-12) | Baseline, 6 weeks (post-intervention), 12 weeks (follow-up)
  The Medical Outcomes Study (MOS) SF-12 is a valid and reliable self-administered questionnaire assessing health-related quality-of-life and change in health status. The SF-12 consists of 12-items that measure eight health domains of physical and mental health. The items use either 2- or 3 point, or 5- or 6-point Likert-scales and a summary score reflecting physical and mental health is calculated using weighted means of the domains to asses perceived change in QOL and health. Scores range from 0-30. Higher scores reflect greater QOL and health.
Work and Social Adjustment Scale (WSAS) | Baseline, 6 weeks (post-intervention), 12 weeks (follow-up)
  The WSAS is a validated and reliable brief, 5-item global measure of functional impairment for adults with clinical symptoms of mental illness. Items are scored on a 9-point Likert-scale ranging from 0 = Not at All, 2 = Slightly, 4 = Definitely, 6 = Markedly, 8 = Very Severely. Total WSAS score ranges from 0 to 40 with 0-9 = low impairment (subclinical populations), 10-19 = moderate impairment (less severe), and scores > 20 suggesting severe impairment or worse psychopathology.
Probabilistic instrumental learning task (PILT) | Baseline, 6 weeks (post-intervention), 12 weeks (follow-up)
  The PILT task assesses reward learning via computer task. Participants make decisions between four sets of two abstract choice symbols each associated with a fixed reward probability. Two pairs of symbols displayed on a computer screen for 4s: One pair is associated with "win" outcomes (win £ or no change) and the other with loss outcomes (lose £ or no change). Each symbol within the pair has reciprocal probabilities (70% or 30%) of either outcome occurring (win or loss). Participants complete sixty trials (30 win, 30 loss) and receive outcome feedback (win or loss) after each trial. Participants use the outcome feedback to gradually learn the symbol-outcome win/loss associations to consistently choose the symbol with the high-probability win and avoid the symbol with the high-probability loss. Outcomes assessed include end total £, amount £ won, amount £ lost, reward vs. loss trials, and number of choice switches.
Cortisol Awakening Response (CAR; Saliva) | Baseline, 6 weeks (post-intervention)
  The CAR test measures circadian cortisol rhythm within the first hour after waking from sleep. The test includes 4 small tubes for collecting saliva samples upon waking, 30-minutes after, 45-minutes after, and 60-minutes after to assess the response of the HPA axis by measuring fluctuating cortisol levels. The CAR has emerged as a marker of hypothalamic-pituitary-adrenocortical (HPA) axis function and is related to stress, affective disorders and physical health risk.
Gut microbiome (Stool) | Baseline, 6 weeks (post-intervention)
  The gut microbiome stool test will measure changes in microbiome compositions before and after the intervention. A test kit will be sent to participants to collect a stool sample. Extracted faecal information will be sequenced to obtain a global representation of the microbiome compositions, and Alpha diversity will be measured using Observed Species, Whole Tree Phylogeny, and Shannon and Simpson indices.

OTHER OUTCOMES:
Weight | Baseline, 6 weeks (post-intervention), 12 weeks (follow-up)
  Changes in body weight will be monitored and assessed using study-provided weight scales if participants do not have one. The intervention is not aiming to reduce body weight, but weight will be monitored to ensure ketogenic diet intake is isoenergetic.

CONTACTS AND LOCATIONS:
Overall Officials: Min Gao, PhD, Principal Investigator — University of Oxford; Megan Kirk Chang, PhD, Principal Investigator — University of Oxford; Paul Aveyard, PhD, FRCGP, Study Director — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol, statistical analysis plan, and individual participant data (IPD) that underlie the results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after publication in a peer-reviewed journal for a period of up to 12-months.
Access Criteria: Please contact the primary investigators listed on this trial registration for access.

REFERENCES:
- [Background] Ali S, Rhodes L, Moreea O, McMillan D, Gilbody S, Leach C, Lucock M, Lutz W, Delgadillo J. How durable is the effect of low intensity CBT for depression and anxiety? Remission and relapse in a longitudinal cohort study. Behav Res Ther. 2017 Jul;94:1-8. doi: 10.1016/j.brat.2017.04.006. Epub 2017 Apr 18. PMID 28437680
- [Background] Chesney E, Goodwin GM, Fazel S. Risks of all-cause and suicide mortality in mental disorders: a meta-review. World Psychiatry. 2014 Jun;13(2):153-60. doi: 10.1002/wps.20128. PMID 24890068
- [Background] Johnson CF, Macdonald HJ, Atkinson P, Buchanan AI, Downes N, Dougall N. Reviewing long-term antidepressants can reduce drug burden: a prospective observational cohort study. Br J Gen Pract. 2012 Nov;62(604):e773-9. doi: 10.3399/bjgp12X658304. PMID 23211181
- [Background] Martin K, Jackson CF, Levy RG, Cooper PN. Ketogenic diet and other dietary treatments for epilepsy. Cochrane Database Syst Rev. 2016 Feb 9;2:CD001903. doi: 10.1002/14651858.CD001903.pub3. PMID 26859528
- [Background] Garcia-Rodriguez D, Gimenez-Cassina A. Ketone Bodies in the Brain Beyond Fuel Metabolism: From Excitability to Gene Expression and Cell Signaling. Front Mol Neurosci. 2021 Aug 27;14:732120. doi: 10.3389/fnmol.2021.732120. eCollection 2021. PMID 34512261
- [Background] Zarnowski T, Choragiewicz T, Tulidowicz-Bielak M, Thaler S, Rejdak R, Zarnowski I, Turski WA, Gasior M. Ketogenic diet increases concentrations of kynurenic acid in discrete brain structures of young and adult rats. J Neural Transm (Vienna). 2012 Jun;119(6):679-84. doi: 10.1007/s00702-011-0750-2. Epub 2011 Dec 27. PMID 22200857
- [Background] Page CE, Coutellier L. Prefrontal excitatory/inhibitory balance in stress and emotional disorders: Evidence for over-inhibition. Neurosci Biobehav Rev. 2019 Oct;105:39-51. doi: 10.1016/j.neubiorev.2019.07.024. Epub 2019 Aug 1. PMID 31377218
- [Background] Duman RS, Sanacora G, Krystal JH. Altered Connectivity in Depression: GABA and Glutamate Neurotransmitter Deficits and Reversal by Novel Treatments. Neuron. 2019 Apr 3;102(1):75-90. doi: 10.1016/j.neuron.2019.03.013. PMID 30946828
- [Background] Yudkoff M, Daikhin Y, Nissim I, Horyn O, Lazarow A, Luhovyy B, Wehrli S, Nissim I. Response of brain amino acid metabolism to ketosis. Neurochem Int. 2005 Jul;47(1-2):119-28. doi: 10.1016/j.neuint.2005.04.014. PMID 15888376
- [Background] Duking T, Spieth L, Berghoff SA, Piepkorn L, Schmidke AM, Mitkovski M, Kannaiyan N, Hosang L, Scholz P, Shaib AH, Schneider LV, Hesse D, Ruhwedel T, Sun T, Linhoff L, Trevisiol A, Kohler S, Pastor AM, Misgeld T, Sereda M, Hassouna I, Rossner MJ, Odoardi F, Ischebeck T, de Hoz L, Hirrlinger J, Jahn O, Saher G. Ketogenic diet uncovers differential metabolic plasticity of brain cells. Sci Adv. 2022 Sep 16;8(37):eabo7639. doi: 10.1126/sciadv.abo7639. Epub 2022 Sep 16. PMID 36112685
- [Background] Guan YF, Huang GB, Xu MD, Gao F, Lin S, Huang J, Wang J, Li YQ, Wu CH, Yao S, Wang Y, Zhang YL, Teoh JP, Xuan A, Sun XD. Anti-depression effects of ketogenic diet are mediated via the restoration of microglial activation and neuronal excitability in the lateral habenula. Brain Behav Immun. 2020 Aug;88:748-762. doi: 10.1016/j.bbi.2020.05.032. Epub 2020 May 12. PMID 32413556
- [Background] Brietzke E, Mansur RB, Subramaniapillai M, Balanza-Martinez V, Vinberg M, Gonzalez-Pinto A, Rosenblat JD, Ho R, McIntyre RS. Ketogenic diet as a metabolic therapy for mood disorders: Evidence and developments. Neurosci Biobehav Rev. 2018 Nov;94:11-16. doi: 10.1016/j.neubiorev.2018.07.020. Epub 2018 Jul 31. PMID 30075165
- [Background] Fattal O, Budur K, Vaughan AJ, Franco K. Review of the literature on major mental disorders in adult patients with mitochondrial diseases. Psychosomatics. 2006 Jan-Feb;47(1):1-7. doi: 10.1176/appi.psy.47.1.1. PMID 16384802
- [Background] Yarar-Fisher C, Li J, Womack ED, Alharbi A, Seira O, Kolehmainen KL, Plunet WT, Alaeiilkhchi N, Tetzlaff W. Ketogenic regimens for acute neurotraumatic events. Curr Opin Biotechnol. 2021 Aug;70:68-74. doi: 10.1016/j.copbio.2020.12.009. Epub 2021 Jan 11. PMID 33445134
- [Background] Puchowicz MA, Xu K, Sun X, Ivy A, Emancipator D, LaManna JC. Diet-induced ketosis increases capillary density without altered blood flow in rat brain. Am J Physiol Endocrinol Metab. 2007 Jun;292(6):E1607-15. doi: 10.1152/ajpendo.00512.2006. Epub 2007 Feb 6. PMID 17284577
- [Background] Jarrett SG, Milder JB, Liang LP, Patel M. The ketogenic diet increases mitochondrial glutathione levels. J Neurochem. 2008 Aug;106(3):1044-51. doi: 10.1111/j.1471-4159.2008.05460.x. Epub 2008 May 5. PMID 18466343
- [Background] Villa RF, Ferrari F, Bagini L, Gorini A, Brunello N, Tascedda F. Mitochondrial energy metabolism of rat hippocampus after treatment with the antidepressants desipramine and fluoxetine. Neuropharmacology. 2017 Jul 15;121:30-38. doi: 10.1016/j.neuropharm.2017.04.025. Epub 2017 Apr 18. PMID 28431972
- [Background] Guarnotta V, Emanuele F, Amodei R, Giordano C. Very Low-Calorie Ketogenic Diet: A Potential Application in the Treatment of Hypercortisolism Comorbidities. Nutrients. 2022 Jun 9;14(12):2388. doi: 10.3390/nu14122388. PMID 35745118
- [Background] Ebbeling CB, Feldman HA, Klein GL, Wong JMW, Bielak L, Steltz SK, Luoto PK, Wolfe RR, Wong WW, Ludwig DS. Effects of a low carbohydrate diet on energy expenditure during weight loss maintenance: randomized trial. BMJ. 2018 Nov 14;363:k4583. doi: 10.1136/bmj.k4583. PMID 30429127
- [Background] Karkkainen O, Farokhnia M, Klavus A, Auriola S, Lehtonen M, Deschaine SL, Piacentino D, Abshire KM, Jackson SN, Leggio L. Effect of intravenous ghrelin administration, combined with alcohol, on circulating metabolome in heavy drinking individuals with alcohol use disorder. Alcohol Clin Exp Res. 2021 Nov;45(11):2207-2216. doi: 10.1111/acer.14719. Epub 2021 Sep 30. PMID 34590334
- [Background] Attaye I, van Oppenraaij S, Warmbrunn MV, Nieuwdorp M. The Role of the Gut Microbiota on the Beneficial Effects of Ketogenic Diets. Nutrients. 2021 Dec 31;14(1):191. doi: 10.3390/nu14010191. PMID 35011071
- [Background] Bough KJ, Wetherington J, Hassel B, Pare JF, Gawryluk JW, Greene JG, Shaw R, Smith Y, Geiger JD, Dingledine RJ. Mitochondrial biogenesis in the anticonvulsant mechanism of the ketogenic diet. Ann Neurol. 2006 Aug;60(2):223-35. doi: 10.1002/ana.20899. PMID 16807920
- [Background] Hallbook T, Ji S, Maudsley S, Martin B. The effects of the ketogenic diet on behavior and cognition. Epilepsy Res. 2012 Jul;100(3):304-9. doi: 10.1016/j.eplepsyres.2011.04.017. Epub 2011 Aug 27. PMID 21872440
- [Background] van Berkel AA, IJff DM, Verkuyl JM. Cognitive benefits of the ketogenic diet in patients with epilepsy: A systematic overview. Epilepsy Behav. 2018 Oct;87:69-77. doi: 10.1016/j.yebeh.2018.06.004. Epub 2018 Aug 31. PMID 30173019
- [Background] Dietch DM, Kerr-Gaffney J, Hockey M, Marx W, Ruusunen A, Young AH, Berk M, Mondelli V. Efficacy of low carbohydrate and ketogenic diets in treating mood and anxiety disorders: systematic review and implications for clinical practice. BJPsych Open. 2023 Apr 17;9(3):e70. doi: 10.1192/bjo.2023.36. PMID 37066662
- [Background] Cuijpers P, Karyotaki E, Weitz E, Andersson G, Hollon SD, van Straten A. The effects of psychotherapies for major depression in adults on remission, recovery and improvement: a meta-analysis. J Affect Disord. 2014 Apr;159:118-26. doi: 10.1016/j.jad.2014.02.026. Epub 2014 Feb 24. PMID 24679399
- [Background] Khan A, Brown WA. Antidepressants versus placebo in major depression: an overview. World Psychiatry. 2015 Oct;14(3):294-300. doi: 10.1002/wps.20241. PMID 26407778
- [Background] Cummergen K, Hannah L, Jopling L, Cameron R, Walsh C, Perez J. What outcomes matter to service users who experience persistent depression: A mixed-method narrative review and synthesis. Journal of Affective Disorders Reports 2022; 10: 100431.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Lam RW, Lamy FX, Danchenko N, Yarlas A, White MK, Rive B, Saragoussi D. Psychometric validation of the Perceived Deficits Questionnaire-Depression (PDQ-D) instrument in US and UK respondents with major depressive disorder. Neuropsychiatr Dis Treat. 2018 Oct 29;14:2861-2877. doi: 10.2147/NDT.S175188. eCollection 2018. PMID 30464471
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Walsh AEL, Browning M, Drevets WC, Furey M, Harmer CJ. Dissociable temporal effects of bupropion on behavioural measures of emotional and reward processing in depression. Philos Trans R Soc Lond B Biol Sci. 2018 Mar 19;373(1742):20170030. doi: 10.1098/rstb.2017.0030. PMID 29352029
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Miletic S, Boag RJ, Trutti AC, Stevenson N, Forstmann BU, Heathcote A. A new model of decision processing in instrumental learning tasks. Elife. 2021 Jan 27;10:e63055. doi: 10.7554/eLife.63055. PMID 33501916
- [Background] Mordor Intelligence LLC. Global Ketogenic Diet Food Market - Growth, Trends and Forecast (2019 - 2024). 2019. https://www.reportlinker.com/p05790924/Global-Ketogenic-Diet-Food-Market-Growth-Trends-and-Forecast.html#:~:text=The%20global%20ketogenic%20diet%20food,and%20aiding%20in%20weight%2Dloss.
- [Derived] Gao M, Kirk M, Knight H, Lash E, Michalopoulou M, Guess N, Stevens R, Browning M, Weich S, Burnet PWJ, Jebb SA, Aveyard P. A Ketogenic Diet for Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2026 Feb 4:e254431. doi: 10.1001/jamapsychiatry.2025.4431. Online ahead of print. PMID 41637092